CLINICAL TRIAL: NCT05443256
Title: Causal Dissociation of Value Contributions to the Reward Positivity
Brief Title: TMS Alteration of the Reward Positivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, James Cavanagh, Associate Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20071
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Anhedonia
MeSH Terms: conditions — Anhedonia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Two separate arms of study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Theta Stim (Experimental): To stimulate fMRI-informed individualized targets in dlPFC to diminish affective modulation of the RewP. Based on our working hypothesis, TMS Figure-8 coil stimulation should diminish affective modulation of RewP amplitude when compared to sham.
  Interventions: Device: Transcranial Magnetic Stimulation
- Sham Stim (Sham Comparator): Sham stimulation. The Reward Positivity should be unaffected.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Figure 8 coil stimulation

SUMMARY:
The aim of this proposal is to demonstrate that stimulation of different brain regions differently affects the electroencephalographic feature known as the Reward Positivity (RewP).

DETAILED DESCRIPTION:
The aim of this proposal is to demonstrate that stimulation of different brain regions differently affects the electroencephalographic feature known as the Reward Positivity (RewP). The RewP is a sensitive and specific biomarker of reward receipt. This proposal will advance a causal test of the hypothesis that there are two major sources of variance that contribute to this brain response: a dorsal midline contribution to information encoding and a ventral midline contribution that is modulated by affect. Together, these findings will reveal how the RewP acts to blend multiple aspects of value together in the service of motivated learning. The objective of this proposal is to gather pilot data to demonstrate the feasibility of using transcranial magnetic stimulation (TMS) to perturb idiosyncratically-defined (fMRI-based) dorsal or ventral targets in order to causally test the hypothesis that these different sources contribute different types of variance to the RewP. TMS double cone deep coil stimulation should diminish +RPE encoding in the RewP when compared to sham. TMS Figure-8 coil stimulation should diminish affective modulation of RewP amplitude when compared to sham.

ELIGIBILITY:
Inclusion Criteria:

• Men or women aged 18-30

Exclusion Criteria:

* Participants unwilling or unable to give informed consent
* Presence of other known medical or psychiatric comorbidity that in the investigator's opinion would compromise participation in the study
* MEG/MRI contraindications
* History of psychosis
* Not fluent in English

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2024-10-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico - Logan hall, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Theta Stim | Sham Stim
Started | 5 | 4
Completed | 4 | 4
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- dlPFC Stimulation: To stimulate fMRI-informed individualized targets in dlPFC to diminish affective modulation of the RewP. Based on our working hypothesis, TMS Figure-8 coil stimulation should diminish affective modulation of RewP amplitude when compared to sham.
  Transcranial Magnetic Stimulation: Figure 8 coil stimulation
- dmPFC Stimulation: To stimulate individualized targets in dmPFC to alter affective modulation of the RewP. Based on our working hypothesis, TMS Deep Cone stimulation should boost learning-related modulation of RewP amplitude when compared to sham.
  Transcranial Magnetic Stimulation: Deep Cone stimulation
- Total: Total of all reporting groups
Arm/Group | dlPFC Stimulation | dmPFC Stimulation | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.75 (5.12) | 29.75 (3.77) | 27.75 (4.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 2 | 5
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Reward Positivity
Description: EEG Amplitude 200-400 ms following reward receipt
Time Frame: During intervention
Measure: Mean (Standard Deviation); unit: femtoteslas
Arm/Group | dlPFC Stimulation | dmPFC Stimulation
Number analyzed (Participants) | 4 | 4
femtoteslas | 2.21 (1.24) | .29 (1.47)

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | dlPFC Stimulation | dmPFC Stimulation
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT05443256/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT05443256/SAP_002.pdf